CLINICAL TRIAL: NCT00668031
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel Design, 2-Arm Study to Investigate the Effect of Aprotinin on Transfusion Requirements and Blood Loss in Patients Undergoing Elective Primary Total Hip Replacement Surgery
Brief Title: Effect of Aprotinin on Transfusion Requirements and Blood Loss in Patients Undergoing Elective Primary Total Hip Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11694
Record Dates: First submitted 2008-04-22; First posted 2008-04-28 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Blood Loss, Surgical
Keywords: Transfusion requirements; Hip replacement surgery; Prevention of blood loss; Bloodloss
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Aprotinin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Trasylol (Aprotinin, BAYA0128)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trasylol (Aprotinin, BAYA0128) — A loading dose IV infusion of 2,000,000 KIU (200 mL) followed by 500,000 KIU (50 mL) IV per hour until the end of surgery of aprotinin using an IV infusion pump
  Arms: Arm 1
Drug: Placebo — A loading dose IV infusion of 2,000,000 KIU (200 mL) followed by 500,000 KIU (50 mL) IV per hour until the end of surgery of of placebo using an IV infusion pump
  Arms: Arm 2

SUMMARY:
The purpose of this study is to assess if aprotinin (BAY A0128), given intravenously during surgery, is safe and can help reduce the amount of bleeding and the need for a blood transfusion during hip replacement surgery. Patients undergoing major surgery are at risk for significant blood loss. Because of this, there is a need for drugs that will help slow the amount of bleeding during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects requiring elective primary total hip replacement surgery
* Documented, signed, dated informed consent obtained prior to any study specific procedures being performed

Exclusion Criteria:

* Subjects with previous exposure to aprotinin in the last 6 months. If the subject has undergone cardiac surgery in the last 6 months, all attempts should be made to ascertain if aprotinin was administered during cardiac surgery. If no records are available, subject should be excluded. If during cardiac surgery in the last 6 months, there is a record of aprotinin administration, subject should be excluded
* Subjects with a known or suspected allergy to aprotinin - Subjects with impaired renal function (serum creatinine > 3.5 mg/dl or 309 micromoles/liter)
* Subjects with a history of bleeding diathesis or known coagulation factor deficiency
* Subjects with failure of a major organ system or any active significant medical illness that in the opinion of the investigator is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study
* Subjects who refuse to receive allogenic blood products for religious or other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2005-02; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Percent of subjects requiring a blood transfusion (predonated blood or packed red blood cells, autologous or allogenic) anytime in the intra-operative or post-operative period (up to the earlier of Day 7 or discharge) | intra-op tp discharge

SECONDARY OUTCOMES:
The percent of subjects receiving an allogenic transfusion of blood or packed red cells during surgery and up to the earlier of Day 7 or discharge. | surgery to discharge
The percent of subjects who did and did not predonate blood receiving an allogenic transfusion of blood or packed red cells during surgery and up to the earlier of Day 7 or discharge. | surgery to discharge
The number of units of blood or packed red cells transfused. There will be analyses for the combination of autologous and allogenic transfusion and for allogenic alone. | surgery to discharge
The number of units of blood or packed red cells transfused per patient requiring transfusion. | surgery to discharge
The estimated blood loss during surgery, drainage (in milliliters) from the operative site in the first six hours post-operatively, and total drainage until removal of drains. | surgery to discharge
The change from preoperative hemoglobin concentration to postoperative hemoglobin concentration (obtained in the morning of postoperative Day 2, or, if transfused earlier, prior to transfusion | pre-operative through day 2
Surgeon's assessment of the degree to which bleeding obscures his/her view of the surgical field, relative to past, similar procedures. | surgery
Changes in blood markers related to inflammation and blood coagulation | surgery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (39):
- United States (27):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - La Jolla, California
  - San Diego, California
  - Aurora, Colorado
  - Farmington, Connecticut
  - Bay Pines, Florida
  - Jacksonville Beach, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Boise, Idaho
  - Indianapolis, Indiana
  - Mooresville, Indiana
  - Iowa City, Iowa
  - Baltimore, Maryland
  - Worcester, Massachusetts
  - Kalamazoo, Michigan
  - Ypsilanti, Michigan
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Bend, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Lubbock, Texas
  - San Antonio, Texas
- Canada (11):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Fredericton, New Brunswick
  - Halifax, Nova Scotia
  - Guelph, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Oshawa, Ontario
  - Richmond Hill, Ontario
  - Québec, Quebec
- San Juan, Puerto Rico